CLINICAL TRIAL: NCT02054767
Title: Anesthetic Efficacy of Articaine, Lidocaine and Mepivacaine in Patients With Irreversible Pulpitis of Mandibular Molar
Brief Title: Anesthetic Efficacy in Irreversible Pulpitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Isabel Peixoto Tortamano, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FDAAA
Record Dates: First submitted 2013-09-03; First posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2013-09

CONDITIONS: Anesthesia
Keywords: articaine; lidocaine; mepivacaine; inferior alveolar nerve block; irreversible pulpitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- lidocaine (Experimental): injections of 3.6 mL of 2% lidocaine with 1:100,000 epinephrine Intervention: inferior alveolar nerve block injection
  Interventions: Drug: Intervention: inferior alveolar nerve block injection
- mepivacaine (Experimental): injections of 3.6 mL of 2% mepivacaine with 1:100,000 epinephrine Intervention: inferior alveolar nerve block injection
  Interventions: Drug: Intervention: inferior alveolar nerve block injection
- articaine (Experimental): injections of 3.6 mL of 4% articaine with 1:100,000 epinephrine Intervention: inferior alveolar nerve block injection
  Interventions: Drug: Intervention: inferior alveolar nerve block injection

INTERVENTIONS:
Drug: Intervention: inferior alveolar nerve block injection — -22 patients received inferior alveolar nerve block injections of 3.6 mL (equivalent to 2 cartridges)

SUMMARY:
The purpose of this study was to compare the anesthetic efficacy of articaine, lidocaine and mepivacaine in patients with irreversible pulpitis of mandibular molar.

DETAILED DESCRIPTION:
Conventional inferior alveolar nerve block (IANB) is the most commonly used technique for achieving pulpal anesthesia in posterior mandibular endodontic procedures. However, IANB has a high failure rate and success rates are even lower when applied for the treatment of mandibular posterior teeth with irreversible pulpitis.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of irreversible pulpitis
* good health
* had at least 1 adjacent tooth plus a healthy canine

Exclusion Criteria:

* took medication could be interacting with any of the anesthetics used

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2010-08; Primary Completion 2012-11 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
pulpal anesthesia | Ten minutes after the inferior alveolar nerve block
  pulpal anesthesia was tested with an electric pulp stimulator

SECONDARY OUTCOMES:
analgesia | the patients were instructed to report any painful sensation at three phases: 1) dentin 2) pulp chamber 3) root canal
  To evaluate the intensity of pain during the pulpectomy a verbal analogic scale was adopted

OTHER OUTCOMES:
lip anesthesia | ten minutes after the inferior alveolar nerve block
  The investigators evaluated the subjective lip anethesia by asking the patient whether his/her lip was numb

CONTACTS AND LOCATIONS:
Overall Officials: Isabel P Tortamano, PhD, Principal Investigator — USão Paulo
Locations (1):
- Emergency Center of the School of Dentistry at the University of São Paulo, São Paulo, São Paulo, Brazil